CLINICAL TRIAL: NCT02615340
Title: Feasibility of Melatonin for Prevention of Delirium in Critically Ill Patients: a Multi-centre, Randomized, Placebo-controlled Study.
Brief Title: Melatonin for Prevention of Delirium in Critically Ill Patients
Acronym: MELLOW-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4000145150
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Delirium
Keywords: delirium; melatonin; pharmacokinetics; feasibility; prevention
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel, patients, and their families will remain blinded. Treatment allocation will only be known to the clinical trials pharmacist, who will perform subject randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enteral melatonin 0.5 mg (Active Comparator): Melatonin 0.5 mg from the 1mg/mL oral suspension qs to 5 mL with Oral Mix SF (sugar-free flavoured suspending vehicle) (final concentration of 0.1 mg/mL; final volume in the oral syringe will be 5 mL)
  Interventions: Drug: Melatonin
- Enteral melatonin 2 mg (Active Comparator): Melatonin 2 mg from the 1mg/mL oral suspension qs to 5 mL with Oral Mix SF (sugar-free flavoured suspending vehicle) (final concentration 0.4 mg/mL; final volume in the oral syringe will be 5 mL)
  Interventions: Drug: Melatonin
- Enteral matched placebo (Placebo Comparator): Melatonin 0 mg qs to 5 mL with Oral Mix SF (sugar-free flavoured suspending vehicle) (final concentration 0 mg/mL; final volume in the oral syringe will be 5 mL)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Study drug will be given at 21:00 - 23:59 daily, starting on the day of enrolment until ICU discharge, death, or up to 14 days, as most critically ill patients are at greatest risk of delirium in the first two weeks of admission. The study medication will be given by mouth (PO or per os) or if needed, via the feeding tube followed by a flush with 20mL water. Doses can be given up to midnight if administration needs to be delayed for procedures or investigations.
  Other Names: N-acetyl-5-methoxytryptamine
  Arms: Enteral melatonin 0.5 mg; Enteral melatonin 2 mg
Drug: Placebo — Study drug will be given at 21:00 - 23:59 daily, starting on the day of enrolment until ICU discharge, death, or up to 14 days, as most critically ill patients are at greatest risk of delirium in the first two weeks of admission. The study medication will be given by mouth (PO or per os) or if needed, via the feeding tube followed by a flush with 20mL water. Doses can be given up to midnight if administration needs to be delayed for procedures or investigations.
  Arms: Enteral matched placebo

SUMMARY:
The purpose of this study is to determine the feasibility of conducting a randomized controlled trial (RCT) with melatonin for prevention of delirium in critically ill adult patients. The investigators hypothesize that melatonin, administered on a scheduled nightly basis during ICU admission, will be efficacious and safe for the prevention of delirium in critically ill adults.

DETAILED DESCRIPTION:
The available evidence indicates melatonin may decrease the incidence of delirium in non-critically ill patient populations; however, trials in the critically ill are lacking. The investigators hypothesize that melatonin, administered on a scheduled nightly basis during ICU admission, will be efficacious and safe for the prevention of delirium in critically ill adults. The null hypothesis is that there is no difference in delirium incidence between placebo and melatonin. Prior to conducting an adequately powered multi-centre, blinded randomized, placebo-controlled trial in critically ill patients, there is a need for a better understanding of melatonin pharmacokinetics (PK) in critically ill patients. This will help to determine appropriate dosing, drug administration issues (specifically protocol adherence), adverse drug effects, and recruitment rates based on inclusion and exclusion criteria.

The specific aim is to conduct a phase II triple blind, placebo-controlled randomized trial comparing two doses of melatonin (low dose = 0.5 mg and high dose = 2.0 mg) to assess the feasibility of a future full-scale RCT. Feasibility of the larger trial will be based on protocol adherence and participant recruitment rates. Data on PK properties of melatonin will be assessed to determine dosing for future studies of melatonin for delirium prevention in the critically ill.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patients ≥18 years of age
2. Anticipated ICU stay of >48 hours
3. Able to receive enteral administration of study drug (i.e. by mouth or any feeding tube = naso- or oro- or percutaneous gastric or post-pyloric feeding tube)
4. Consent to participate.

Exclusion Criteria:

1. ICU admission of >48 hours prior to screening
2. Unable to assess for delirium (e.g. comatose defined as SAS 1 or 2 or either 'No Response' Score A or B on ICDSC, chemically paralyzed with neuromuscular blocking drugs)
3. Screened delirium positive prior to randomization (ICDSC score ≥4 out of 8)
4. Anticipated withdrawal in next 48 hours
5. Known history of severe cognitive or neurodegenerative disease (e.g. dementia, Parkinson's disease) or severe structural brain injury (e.g. traumatic brain injury, intracranial hemorrhage) as the ICDSC assessment tool has not been validated in these patient populations
6. Unable to communicate in English or French (Montreal site)
7. Contraindications to receiving any enteral medication (defined as absolute contraindication to enteral nutrition such as gastrointestinal obstruction, perforation, recent upper GI surgery, no enteral access)
8. Active seizures
9. Known pregnancy
10. Legal blindness
11. Known allergy to melatonin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-10-12 (Estimated); Study Completion 2019-10-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Study adherence | 1 year
  Investigators will calculate protocol adherence as the overall proportion of administered doses in the prescribed dose administration window (between 21:00 and to 23:59 hours) divided by total number of eligible study days.

SECONDARY OUTCOMES:
Feasibility: Trial recruitment | 1 year
  Proportion of ICU patients screened that meet study inclusion criteria, the number of patients excluded and reasons for exclusion, and the consent rate of eligible participants.
Feasibility: Time in motion (minutes) | 1 year
  Research coordinators at each site will capture the amount of time (minutes) taken to screen, consent, and enrol patients, complete study procedures, and collect data.
Pharmacokinetic: Peak melatonin concentration (Cmax) | 24 hours
  Peak melatonin concentration. Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Pharmacokinetic: Time of peak melatonin concentration (Tmax) | 24 hours
  Time of peak melatonin concentration (Tmax). Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Pharmacokinetic: Morning melatonin concentration (C9AM) | 24 hours
  Morning melatonin concentration (C9AM). Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Pharmacokinetic: Melatonin half-life (T½) | 24 hours
  Melatonin half-life (T½). Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Pharmacokinetic: Mean apparent clearance (CL/F) | 24 hours
  Mean apparent clearance (CL/F). Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Pharmacokinetic: Mean apparent volume distribution (V/F) | 24 hours
  Mean apparent volume distribution (V/F). Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Pharmacokinetic: Area under the concentration-time curve (AUC) | 24 hours
  Area under the concentration-time curve (AUC). Plasma melatonin concentrations measured by mass spectrometry. N=5 from each study arm of Mount Sinai Hospital site.
  On study day 1, eight blood samples (4 mL each) will be collected at the following intervals, from the time of first study drug dose to the following morning (time 0, 0.5, 1, 2, 4, 6, 8, 12 hours).
Clinical: Adverse events | 14 days
  Adverse events reported by the participant, family, or treating team. The following potential adverse effects will be collected: morning drowsiness (Sedation Agitation Scale (SAS) score <3 or patient's self report of drowsiness between 07:00h and 12:00h), headache, and vivid dreams.
Clinical: Delirium incidence | 14 days
  Intensive Care Delirium Screening Checklist (ICDSC) administered daily. Delirium defined as an ICDSC score ≥4.
Clinical: Delirium time to onset and duration (days) | 14 days
  Time to onset of first ICDSC score ≥4, and number of days with ICDSC score ≥4.
Clinical: Sleep | 14 days
  Richards Campbell Sleep Questionnaire (RCSQ) administered daily, where possible. Patients with or without the assistance of their nurse will be asked to complete the questions of the RCSQ each morning. Nurses will not complete the RCSQ if the patient is unable to verbalize, as poor correlation has been shown between patient and nursing scores.
Clinical: Duration of mechanical ventilation | ICU admission
  Duration of mechanical ventilation (days)
Clinical: ICU length of stay | ICU admission
  Duration of stay for index ICU admission (days)
Clinical: Hospital length of stay | 1 year
  Duration of stay for admission involving trial enrolment (days)
Clinical: ICU mortality | 1 year
  Number of deaths during index ICU admission
Clinical: Hospital mortality | 1 year
  Number of deaths during hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Burry, PharmD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital du Sacré-Coeur, Montreal, Quebec

REFERENCES:
- [Derived] Burry LD, Williamson DR, Detsky ME, Bernard F, Foster J, Mehta S, Pinto R, Scales DC, Rose L. Low-Dose Melatonin for Prevention of Delirium in Critically Ill Patients: A Multicenter, Randomized, Placebo-Controlled Feasibility Trial. Chest. 2025 May;167(5):1397-1407. doi: 10.1016/j.chest.2024.12.030. Epub 2025 Jan 10. PMID 39800236
- [Derived] Burry L, Scales D, Williamson D, Foster J, Mehta S, Guenette M, Fan E, Detsky M, Azad A, Bernard F, Rose L. Feasibility of melatonin for prevention of delirium in critically ill patients: a protocol for a multicentre, randomised, placebo-controlled study. BMJ Open. 2017 Mar 30;7(3):e015420. doi: 10.1136/bmjopen-2016-015420. PMID 28363933